CLINICAL TRIAL: NCT02447874
Title: Arginine Therapy for the Treatment of Vaso-Occlusive Events in Children With Severe Sickle Cell Disease
Brief Title: Arginine Therapy for the Treatment of Pain in Children With Sickle Cell Disease
Acronym: R34 pK/PD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Claudia R. Morris, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00077736; 1K24AT009893-01 (NIH)
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Standard dose (Experimental): Subjects with sickle cell disease (SCD) and vaso-occlusive painful events (VOE) will be randomized to receive an intravenous (IV) infusion of a standard dose of arginine (100 mg/kg) three times a day for seven days or until discharged from the hospital, whichever occurs first
  Interventions: Drug: Arginine
- Loading dose + standard dose (Experimental): Subjects with sickle cell disease and vaso-occlusive painful events (VOE) will be randomized to receive an intravenous (IV) infusion of an initial loading dose of arginine (200 mg/kg) given over 30 minutes and then receive an intravenous (IV) infusion of a standard dose of arginine (100 mg/kg) three times a day for seven days or until discharged from the hospital, whichever occurs first
  Interventions: Drug: Arginine; Drug: Arginine (Loading)
- Loading dose + continuous infusion (Experimental): Subjects with sickle cell disease and vaso-occlusive painful events (VOE) will be randomized to receive an intravenous (IV) infusion of an initial loading dose of arginine (200 mg/kg) given over 30 minutes and then receive a continuous intravenous (IV) infusion of 300 mg/kg/24hr for 7 days or until discharged from the hospital, whichever occurs first
  Interventions: Drug: Arginine (Loading); Drug: Arginine (Continuous)
- Non-Randomized Loading dose 500 mg/kg + standard dose (Experimental): Arginine will be dispensed intravenously (in the vein) as an initial bolus (loading) arginine dose at 500 mg/kg once, followed by a standard dose of 100mg/kg every 8 hours until discharge or for a total of 21 doses of arginine, whichever comes first.
  Interventions: Drug: Arginine (Loading)
- Non-Randomized Loading dose 300 mg/kg + standard dose (Experimental): Arginine will be dispensed intravenously (in the vein) as an initial bolus (loading) arginine dose at 300 mg/kg once, followed by a standard dose of 100mg/kg every 8 hours until discharge or for a total of 21 doses of arginine, whichever comes first.
  Interventions: Drug: Arginine (Loading)
- Non-Randomized Loading dose 400mg/kg + standard dose (Experimental): Arginine will be dispensed intravenously (in the vein) as an initial bolus (loading) arginine dose at 400 mg/kg once, followed by a standard dose of 100mg/kg every 8 hours until discharge or for a total of 21 doses of arginine, whichever comes first.
  Interventions: Drug: Arginine (Loading)

INTERVENTIONS:
Drug: Arginine — Arginine will be dispensed intravenously (in the vein) in the standard dose of arginine as 100 mg/kg three times a day for seven days or until discharge.
  * Loading dose: 200 mg/kg once
  * Continuous IV: 300 mg/kg/24 hours
  Other Names: Arginine Hydrochloride Injection, R-Gene® 10
  Arms: Loading dose + standard dose; Standard dose
Drug: Arginine (Loading) — Arginine will be dispensed intravenously (in the vein) as an initial bolus (loading) at each specified group dose once, followed by a standard dose of 100mg/kg every 8 hours until discharge or for a total of 21 doses of arginine, whichever comes first.
  Other Names: Arginine Hydrochloride Injection, R-Gene® 10
  Arms: Loading dose + continuous infusion; Loading dose + standard dose; Non-Randomized Loading dose 300 mg/kg + standard dose; Non-Randomized Loading dose 400mg/kg + standard dose; Non-Randomized Loading dose 500 mg/kg + standard dose
Drug: Arginine (Continuous) — Arginine will be dispensed intravenously (in the vein) as a continuous IV infusion of 300 mg/kg/24hr
  Other Names: Arginine Hydrochloride Injection, R-Gene® 10
  Arms: Loading dose + continuous infusion

SUMMARY:
The purpose of this study is to determine whether giving extra arginine to patients with sickle cell disease seeking treatment for vaso-occlusive painful events (VOE) will decrease pain scores, decrease need for pain medications or decrease length of hospital stay or emergency department visit.

DETAILED DESCRIPTION:
Arginine is a simple amino acid that is found in many foods and is part of the proteins in a human's body. Patients with sickle cell disease have low levels of the amino acid arginine and these low levels may be related to pain episodes. Increasing levels of arginine in the blood may lower pain and/or lower the amount of pain medication (like morphine) that is needed to treated them. It may also decrease the amount of time spent in the hospital.

Available data suggest that, L-arginine is a safe & efficacious intervention with narcotic-sparing effects in pediatric SCD patients with VOE. The addition of a higher loading dose to the standard dose or use of a continuous infusion may provide additional clinical benefits by overcoming multiple mechanisms that limit global arginine bioavailability in SCD.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of sickle cell disease--Hemoglobin SS (Hb-SS) or Sβᴼ-thalassemia
* 7-21 years of age
* Weight >= 25kg (55lbs)
* Pain requiring medical care in an acute care setting (emergency department (ED), hospital ward, day hospital, clinic) requiring parenteral opioids, not attributable to non-sickle cell causes.

Exclusion Criteria:

* Decision to discharge home from acute care setting.
* Diagnosis of sickle cell disease with any of the following types: hemoglobin SC disease (HbSC), hemoglobin beta thalassemia (Hb-Beta Thal), hemoglobin SD disease (HbSD), hemoglobin SE disease (HbSE), hemoglobin SO disease (HbSO), hemoglobin AS carrier (Hb AS)
* Hemoglobin less than 5 gm/dL
* Immediate Red cell transfusion anticipated
* Renal dysfunction: Creatinine >1.0 or 2 x baseline
* Mental status or neurological changes
* Acute stroke or clinical concern for stroke
* Pregnancy
* Allergy to arginine
* Previous hospitalization < 7 days
* Use of inhaled nitric oxide, sildenafil or arginine within the last 14 days
* Not an appropriate candidate in the investigator's judgement

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2015-05; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of IV arginine, measured by plasma arginine concentration over time | Day 1 through study completion, an average of up to 7 days
  Total time plasma arginine levels are maintained above the half-saturating concentration (Km) of cationic amino acid transporter protein-1 (CAT-1), which is 150 µM (normal range of extracellular plasma arginine concentration). pK samples will be collected at 6 time-points within 8 hours: prior to arginine treatment (time 0), and at 60, 90, 120 minutes, 4 and 8 hours after the initiation of arginine therapy, and then every 24 hours up to 7 days.
Change in nitric oxide metabolites | Baseline, day 1 through study completion, an average of up to 7 days
  The formation of NO metabolites will be measured by determination of its stable end products in serum; nitrite (NO2-) and nitrate (NO3-). Change in nitric oxide metabolites will be calculated as the difference in metabolites from the time prior to arginine treatment (baseline) to the end of the intervention period.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration -Time Curve (AUC) From Time 0 to the Time of the Last Quantifiable Concentration for Arginine | Day 1
  AUC is derived from drug concentration and time so it gives a measure of how much and how long a drug stays in a body. AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc])
Maximum observed plasma concentration of arginine | Day 1
  Maximum measured concentration of the arginine in plasma
Apparent clearance of arginine | Day 1
  The clearance of a drug measures the rate at which the drug is removed from the body after the dose. Clearance of arginine after intravenous administration on day 1.
Terminal elimination half-life (t1/2) for arginine | Day 1
  Terminal phase elimination half-life (t1/2) is the time required for half of the drug to be eliminated from the plasma.
Change in red blood cell (RBC) arginine | Baseline, day 1 through study completion, an average of up to 7 days
  Change in rbc arginine will be calculated as rbc arginine at the end of arginine administration minus rbc arginine at baseline.
Daily urine arginine | From Day 1 until study completion, an average of up to 7 days
  Total amount of arginine excreted in urine daily
Global arginine bioavailability (GABR) | From enrollment through study completion, an average of up to 7 days
  GABR represents a measure of endothelial function. GABR will be calculated by arginine divided by the sum of ornithine plus citrulline [arginine/(ornithine+citrulline)].
Change in asymmetric dimethylarginine (ADMA) levels | Baseline, day 1 and through study completion, an average of up to 7 days
  ADMA is is a metabolic by-product of continual protein modification processes and interferes with L-arginine in the production of nitric oxide. Change in ADMA levels will be calculated as ADMA levels at the end of arginine administration minus ADMA levels at baseline.
Modeling nitric oxide (NOx) level versus plasma arginine level | From enrollment through study completion, an average of up to 7 days
  Modeling nitric oxide (NOx) level versus plasma arginine level will be measured.
Biomarkers of hemolysis | From enrollment through study completion, an average of up to 7 days
  Biomarkers of hemolysis (lactate dehydrogenase, hemoglobin, reticulocytes, arginase, indirect bilirubin) represent intravascular hemolysis and nitric oxide bioavailability.
Erythrocyte glutathione levels | From enrollment through study completion, an average of up to 7 days
  Erythrocyte glutathione is a biomarker for oxidative stress. It will be measured by using liquid chromatography.
Level of cytokines | From enrollment through study completion, an average of up to 7 days
  Cytokines are biomarkers for inflammation. Cell supernatants will be collected and analyzed for different cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Morris, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare fo Atlanta at Hughes Spalding, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Arthur M. Blank Hospital, Atlanta, Georgia

REFERENCES:
- [Background] Morris CR, Brown LAS, Reynolds M, Dampier CD, Lane PA, Watt A, Kumari P, Harris F, Manoranjithan S, Mendis RD, Figueroa J, Shiva S. Impact of arginine therapy on mitochondrial function in children with sickle cell disease during vaso-occlusive pain. Blood. 2020 Sep 17;136(12):1402-1406. doi: 10.1182/blood.2019003672. PMID 32384147
- [Background] Korman R, Hatabah D, Brown LA, Harris F, Wilkinson H, Rees CA, Bakshi N, Archer DR, Dampier C, Morris CR. Impact of arginine therapy on kyotorphin in children with sickle cell disease and vaso-occlusive pain. Blood Adv. 2024 Jun 25;8(12):3267-3271. doi: 10.1182/bloodadvances.2023012209. PMID 38527291